CLINICAL TRIAL: NCT02264964
Title: Duration and Adverse Events of Non-cuffed Catheter in Patients With Hemodialysis : a Multicenter Prospective Cohort Study
Brief Title: Duration and Adverse Events of Non-cuffed Catheter in Patients With Hemodialysis
Acronym: DACAPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director, Division of Nephrology, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CZHKI-HDVA-002
Record Dates: First submitted 2014-09-23; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Central Venous Catheterization; Inadequate Hemodialysis Blood Flow; Venous Stenosis; Venous Thrombosis; Infection Due to Central Venous Catheter; Central Venous Catheter Thrombosis
Keywords: Hemodialysis; End-Stage Kidney Disease; Central Venous Catheterization; Digital Subtraction Angiography
MeSH Terms: conditions — Venous Thrombosis; Upper Extremity Deep Vein Thrombosis; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- internal jugular vein catheterization (Experimental): 900 patients will be received temporary central vena catheterization in right internal jugular vein with non-cuff GamCath® catheter.They will undergo AVF creation.
  Interventions: Device: GamCath®; Procedure: Arteriovenous fistula creation
- femoral vein catheterization (Experimental): 500 patients will be received temporary central vena catheterization in femoral vein with non-cuff GamCath® catheter, which are unsuitable for right internal jugular vein catheterization.They will undergo AVF creation.
  Interventions: Device: GamCath®; Procedure: Arteriovenous fistula creation

INTERVENTIONS:
Device: GamCath® — Using non-cuff GamCath® catheter in patients with chronic renal failure requiring hemodialysis to building short-term vascular access in femoral vein.
  Other Names: radiopaque catheter(11F) polyurethane
  Arms: femoral vein catheterization
Procedure: Arteriovenous fistula creation — 500 patients will undergo AVF creation in either arm for femoral vein catheterization group.
  Other Names: Arteriovenous fistulization; AVF creation
  Arms: femoral vein catheterization
Device: GamCath® — Using non-cuff GamCath® catheter in patients with chronic renal failure requiring hemodialysis to building short-term vascular access in right internal jugular vein.
  Other Names: radiopaque catheter(11F) polyurethane with curved extension lines
  Arms: internal jugular vein catheterization
Procedure: Arteriovenous fistula creation — 900 patients will undergo AVF creation in left arm for internal jugular vein catheterization group.
  Other Names: Arteriovenous fistulization; AVF creation
  Arms: internal jugular vein catheterization

SUMMARY:
The duration and adverse events of non-cuffed catheter in patients with hemodialysis will be investigated by multicenter prospective cohort. Totally, 1,400 patients with chronic renal failure requiring hemodialysis will be enrolled. 900 patients will be given right internal jugular catheterization, and the other 500 patients unsuitable for right internal jugular catheterization will receive femoral catheterizations. Every patient will be followed-up for six months. During following-up period, the duration time and adverse events of non-cuffed catheter will be recorded in details, including inadequate hemodialysis blood flow, venous stenosis, venous thrombosis, infection, catheter thrombosis and so on. The central vein will be evaluated by CT Angiography to identify its stenosis at last visit after 6 months. This multicentre trial will provide evidence to develop guideline for duration time of using non-cuffed catheter.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure requiring hemodialysis.
* No medical history of central vena catheterization.
* Maintenance hemodialysis after central vena catheterization.
* Signed informed consent.

Exclusion Criteria:

* Had been performed central venous puncture or catheterization before.
* Can not use heparin.
* Refused to sign the informed consent.
* Advanced cancer patients.
* With or will take arteriovenous fistula surgery in right arm.
* Other inappropriate situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bloodstream infection due to central venous catheter | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
Central venous catheter exit site infection | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
Inadequate hemodialysis blood flow | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
Central venous catheter thrombosis | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
venous thrombosis | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
venous stenosis | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.
Duration time of non-cuff catheter | up to 3 months
  Participants will be followed-up during non-cuffed catheter retention, an expected up to 3 months.

SECONDARY OUTCOMES:
Long term occurrence of venous stenosis | 6 months
  CT Angiography for punctured vein will be performed to identify vein stenosis in last visit after 6 months.
Effects on ECG | From baseline to 6months
  ECG will be performed in preoperative, postoperative, catheter removal and last visit after 6 months.
Safety Evaluation | From baseline to 6months
  adverse event or serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, master, Principal Investigator — Division of Nephrology, Shanghai ChangZheng Hospital